CLINICAL TRIAL: NCT05409183
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Clinical Study to Assess the Effectiveness of CRD-740 in Subjects With Chronic Heart Failure (CARDINAL-HF)
Brief Title: Effectiveness of CRD-740 in Heart Failure
Acronym: CARDINAL-HF
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Part A of the study was successfully concluded. Part B of the study was not conducted in favor of redesigned new studies.
Sponsor: Cardurion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRD-740-201
Record Dates: First submitted 2022-06-03; First posted 2022-06-08 (Actual); Results first posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-11

CONDITIONS: Heart Failure; Heart Failure With Reduced Ejection Fraction; Heart Failure With Preserved Ejection Fraction; Cardiovascular Diseases; Heart Diseases
Keywords: PDE9; Heart Failure; CRD-740; HFpEF; HFrEF
MeSH Terms: conditions — Heart Failure; Cardiovascular Diseases; Heart Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CRD-740 (Experimental): Part A: Participants in Part A randomly assigned to this arm will take CRD-740 at two ascending dose levels over 12 weeks.
  Interventions: Drug: CRD-740
- Placebo (Placebo Comparator): Part A: Participants in Part A randomly assigned to this arm will take placebo at two ascending dose levels over 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CRD-740 — Tablets administered orally.
  Arms: CRD-740
Drug: Placebo — Tablets administered orally.
  Arms: Placebo

SUMMARY:
This is a study evaluating the effectiveness of CRD-740 in patients with either Heart Failure with Reduced Ejection Fraction (HFrEF) or Heart Failure with Preserved Ejection Fraction (HFpEF) after 12 weeks of treatment. The primary objective in Part A is to assess the effect of CRD-740 compared to placebo in plasma cGMP at Week 4 in HFrEF.

Part B of the study was not conducted in favor of redesigned new studies.

ELIGIBILITY:
Inclusion Criteria:

1. Males or Females ≥18 years of age, at screening.
2. Diagnosis of clinical heart failure syndrome, New York Heart Association functional class II - III for at least 6 months prior to screening
3. For Part A:

   * Ejection Fraction ≤40% by echocardiography at screening.
   * NT-proBNP level ≥600 pg/ml at screening. Subjects with atrial fibrillation or flutter at screening are required to have an NT-proBNP level of ≥1000 pg/mL at screening.

5. Stable doses of guideline-directed heart failure therapy for a minimum of 4 weeks prior to screening that has been individually optimized according to standard practice guidelines and no addition of guideline-directed heart failure therapy within 3 months of screening.

Exclusion Criteria:

2. Recent HF exacerbation defined by hospitalization or requirement for intravenous diuretics within 60 days of screening.

3. Subjects with planned interventions (e.g., percutaneous coronary intervention, devices) etc. occurring during their involvement in this study.

4. Acute coronary syndrome, stroke, transient ischemic attack, cardiac, carotid or other major cardiovascular surgery or carotid angioplasty within 60 days of screening.

5. Subjects with clinical suspicion of infiltrative cardiomyopathy (e.g., amyloid, sarcoid), hypertrophic cardiomyopathy (obstructive or non-obstructive), or HF secondary to severe valvular disease, active myocarditis, active pericarditis, or clinically significant congenital heart disease.

6. Prior or planned orthotopic heart transplantation.

7. Presence of or plan for mechanical circulatory support.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-05-26 (Actual); Primary Completion 2023-05-02 (Actual); Study Completion 2023-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard Surks, MD, Study Director — Chief Medical and Scientific Officer
Locations (32):
- United States (16):
  - Cardurion Investigative Site, Alexander City, Alabama
  - Cardurion Investigative Site, Birmingham, Alabama
  - Cardurion Investigative Site, Fairhope, Alabama
  - Cardurion Investigative Site, Torrance, California
  - Cardurion Investigative Site, Hialeah, Florida
  - Cardurion Investigative Site, Miami, Florida
  - Cardurion Investigative Site, Naples, Florida
  - Cardurion Investigative Site, Tampa, Florida
  - Cardurion Investigative Site, Atlanta, Georgia
  - Cardurion Investigative Site, Hazel Crest, Illinois
  - Cardurion Investigative Site, Alexandria, Louisiana
  - Cardurion Investigative Site, Minneapolis, Minnesota
  - Cardurion Investigative Site, Greensboro, North Carolina
  - Cardurion Investigative Site, Tullahoma, Tennessee
  - Cardurion Investigative Site, Allen, Texas
  - Cardurion Investigative Site, Norfolk, Virginia
- Cardurion Investigative Site, Winnepeg, Manitoba, Canada
- Israel (6):
  - Cardurion Investigative Site, Ashkelon
  - Cardurion Investigative Site, Be’er Ya‘aqov
  - Cardurion Investigative Site, Haifa
  - Cardurion Investigative Site, Nahariya
  - Cardurion Investigative Site, Rehovot
  - Cardurion Investigative Site, Tiberias
- United Kingdom (9):
  - Cardurion Investigative Site, High Wycombe, Buckinghamshire
  - Cardurion Investigative Site, Airdrie, Lanarkshire
  - Cardurion Investigative Site, Isleworth, Middlesex
  - Cardurion Investigative Site, Clydebank
  - Cardurion Investigative Site, Dundee
  - Cardurion Investigative Site, Glasgow
  - Cardurion Investigative Site, Harrow
  - Cardurion Investigative Site, Newcastle upon Tyne
  - Cardurion Investigative Site, Stockton-on-Tees

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Udelson JE, Belohlavek J, Dukat A, Ezekowitz J, Goland S, Merkely B, O'Meara E, Petrie MC, Ponikowski P, Senni M, Tokmakova M, Vardeny O, Claggett B, Moore E, Savard M, McKellar H, Surks HK, Solomon SD, McMurray JJV. Phase 2, Randomized, Double-Blind, Placebo-Controlled Study of CRD-740, a PDE9 Inhibitor, in Chronic Heart Failure. JACC Heart Fail. 2026 Jan;14(1):102706. doi: 10.1016/j.jchf.2025.102706. Epub 2025 Oct 31. PMID 41171251

RESULTS

PARTICIPANT FLOW:
Groups:
- CRD-740: Part A: Participants in Part A randomly assigned to this arm will take CRD-740 at two ascending dose levels over 12 weeks.
  CRD-740: Tablets administered orally.
  Part B of the study was not conducted in favor of redesigned new studies.
- Placebo: Part A: Participants in Part A randomly assigned to this arm will take placebo at two ascending dose levels over 12 weeks.
  Placebo: Tablets administered orally.
  Part B of the study was not conducted in favor of redesigned new studies.
Period: Period 1
Arm/Group | CRD-740 | Placebo
Started | 40 | 20
Completed | 40 | 20
Not Completed | 0 | 0
Period: Period 2
Arm/Group | CRD-740 | Placebo
Started | 40 | 20
Completed | 38 | 19
Not Completed | 2 | 1
Period: Period 3
Arm/Group | CRD-740 | Placebo
Started | 38 | 19
Completed | 36 | 19
Not Completed | 2 | 0
Period: Complete Study
Arm/Group | CRD-740 | Placebo
Started | 40 | 20
Completed | 36 | 18
Not Completed | 4 | 2
Not completed — Adverse Event | 1 | 2
Not completed — Withdrawal by Subject | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CRD-740 | Placebo | Total
Number analyzed (Participants) | 40 | 20 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 9 | 26
  >=65 years | 23 | 11 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.4 (12.70) | 65.6 (13.16) | 67.4 (12.81)
Age, Customized [Median (Full Range); unit: years]
  Median Age | 70.5 [43 to 88] | 66.0 [36 to 87] | 69.0 [36 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 35 | 16 | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 2 | 6
  Not Hispanic or Latino | 36 | 18 | 54
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 4 | 13
  White | 29 | 15 | 44
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 27 | 13 | 40
  United Kingdom | 8 | 4 | 12
  Israel | 5 | 3 | 8
Mean Height (cm) at Baseline [Mean (Standard Deviation); unit: cm] | 175.6 (10.20) | 172.5 (10.65) | 174.6 (10.36)
Median Height (cm) at Baseline [Median (Full Range); unit: cm] | 175.0 [150 to 203] | 170.8 [157 to 195] | 173.4 [150 to 203]
Reproductive System Findings Test (Female only), n (%) [Count of Participants; unit: Participants] — Population: Female population only
  Participants
    Childbearing Potential: number analyzed (Participants) | 5 | 4 | 9
    Childbearing Potential | 2 | 0 | 2
    Menopause Status: number analyzed (Participants) | 5 | 4 | 9
    Menopause Status | 3 | 4 | 7
Mean Weight (kg) at Baseline [Mean (Standard Deviation); unit: kg] | 97.27 (37.582) | 84.07 (16.932) | 92.87 (32.639)
Median Weight (kg) at Baseline [Median (Full Range); unit: kg] | 87.65 [51.3 to 255.4] | 81.00 [65.0 to 128.1] | 85.55 [51.3 to 255.4]
Mean Body Mass Index (kg/m2) at Baseline [Mean (Standard Deviation); unit: body weight (kg)/ height (m2)] | 31.41 (11.483) | 28.38 (5.953) | 30.40 (10.032)
Median Body Mass Index (kg/m2) at Baseline [Median (Full Range); unit: body weight (kg)/ height (m2)] | 28.92 [18.4 to 83.4] | 26.72 [20.8 to 44.8] | 27.89 [18.4 to 83.4]
Echocardiogram performed during screening [Count of Participants; unit: Participants]
  Yes | 40 | 20 | 60
  No | 0 | 0 | 0
EF group [Count of Participants; unit: Participants]
  EF ≤ 40% | 40 | 20 | 60
  EF > 40% | 0 | 0 | 0
Mean EF (%) for rEF (≤40%) subjects [Mean (Standard Deviation); unit: percent] | 29.16 (7.191) | 26.91 (6.181) | 28.41 (6.901)
Median EF (%) for rEF (≤40%) subjects [Median (Full Range); unit: percent] | 26.50 [15.7 to 40.0] | 25.00 [20.0 to 40.0] | 25.00 [15.7 to 40.0]

OUTCOME MEASURES:

1. Primary Outcome: Part A: The Mean Change From Baseline (Day 1) in Plasma cGMP at Week 4.
Description: Efficacy: To assess the effect of CRD-740 compared to placebo in plasma cGMP at Week 4 in subjects with CHFrEF.
Time Frame: Baseline to Week 4
Population: The modified Intention to Treat (mITT) Population will consist of all randomized subjects who received at least one dose of CRD-740 or placebo. Subjects will be analyzed according to their randomized treatment, regardless of actual treatment received, treatment compliance, or treatment duration.
Measure: Mean (Standard Deviation); unit: AUC 0-6hr (hr*nmol/L)
Arm/Group | CRD-740 | Placebo
Number analyzed (Participants) | 30 | 15
AUC 0-6hr (hr*nmol/L) | 19.139 (26.9007) | -8.822 (31.3357)
Statistical Analysis 1: Comparison: CRD-740 vs Placebo; Test type: Other; p = 0.0032, ANCOVA; LS Mean of Treatment Difference = 26.473, 95% CI 2-sided [7.847 to 45.099], Standard Error of Mean 9.2160

ADVERSE EVENTS:
Time Frame: Through week 12 plus a 4-week follow-up period.
Description: For Part A, the primary safety analysis was performed by reporting the exposure-adjusted incidence rates in subject-years for AEs and SAEs defined as the number of subjects with that particular AE or SAE within an SOC or PT during the relevant period divided by the sum of the at-risk times.
Groups:
- Period 1: CRD-740: CRD-740 10 mg was administered BID to randomly assigned participants in this period from Day 1 through Day 14.
- Period 1: Placebo: CRD-740 10 mg matching placebo was administered BID to randomly assigned participants in this period from Day 1 through Day 14.
- Period 2: CRD-740: CRD-740 25 mg was administered BID to randomly assigned participants in this period from Day 15 through Day 28.
- Period 2: Placebo: CRD-740 25 mg matching placebo was administered BID to randomly assigned participants in this period from Day 15 through Day 28.
- Period 3: CRD-740: CRD-740 25 mg was administered BID to randomly assigned participants in this period from Day 29 through Day 84.
- Period 3: Placebo: CRD-740 25 mg matching placebo was administered BID to randomly assigned participants in this period from Day 29 through Day 84.
- Overall CRD-740: Part A: Participants in Part A randomly assigned to this arm will take CRD-740 at two ascending dose levels over 12 weeks plus a 4-week follow-up period.
  CRD-740: Tablets administered orally.
  Part B of the study was not conducted in favor of redesigned new studies.
- Overall Placebo: Part A: Participants in Part A randomly assigned to this arm will take placebo at two ascending dose levels over 12 weeks plus a 4-week follow-up period.
  Placebo: Tablets administered orally.
  Part B of the study was not conducted in favor of redesigned new studies.
Arm/Group | Period 1: CRD-740 | Period 1: Placebo | Period 2: CRD-740 | Period 2: Placebo | Period 3: CRD-740 | Period 3: Placebo | Overall CRD-740 | Overall Placebo
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/20 | 0/38 | 0/19 | 0/36 | 0/19 | 0/40 | 0/20
Serious Adverse Events (participants affected / at risk) | 1/40 | 0/20 | 1/38 | 0/19 | 0/36 | 1/19 | 3/40 | 3/20
Other Adverse Events (participants affected / at risk) | 1/40 | 1/20 | 3/38 | 1/19 | 4/36 | 1/19 | 5/40 | 3/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Period 1: CRD-740 (N=40) | Period 1: Placebo (N=20) | Period 2: CRD-740 (N=38) | Period 2: Placebo (N=19) | Period 3: CRD-740 (N=36) | Period 3: Placebo (N=19) | Overall CRD-740 (N=40) | Overall Placebo (N=20)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal mass (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Period 1: CRD-740 (N=40) | Period 1: Placebo (N=20) | Period 2: CRD-740 (N=38) | Period 2: Placebo (N=19) | Period 3: CRD-740 (N=36) | Period 3: Placebo (N=19) | Overall CRD-740 (N=40) | Overall Placebo (N=20)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness postural (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Scleritis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 1 (4) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
This study was planned to have been conducted in 2 parts: Part A and Part B. Part A was a dose ranging study in a group of subjects with CHFrEF. Part B was planned to be a proof-of-concept study in subjects with either CHFrEF or CHFpEF. Part B of the study was not conducted in favor of redesigned new studies.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-08-10): https://cdn.clinicaltrials.gov/large-docs/83/NCT05409183/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-17): https://cdn.clinicaltrials.gov/large-docs/83/NCT05409183/SAP_001.pdf